CLINICAL TRIAL: NCT06686316
Title: Effects of a 6-week Hypoxia-hyperoxia Exposure Protocol on Sedentary Older Adults on Heart Rate Variability, Blood Pressure, Respiratory Muscle Strength, Pulmonary Function, Inflammatory Biomarkers and Arterial Oxygen Saturation, a Randomized Double-blind Placebo-controlled Clinical Trial
Brief Title: Effects of Intermittent Hypoxia-Hyperoxia in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sierra Varona SL (Other)
Collaborators: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 016
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Sedentary Behavior; Frailty; Older Adults
Keywords: hypoxic training; elderly; heart rate variability
MeSH Terms: conditions — Sedentary Behavior; Frailty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The EG (Experimental Group) will undergo a 6-week intervention protocol with three weekly sessions (Monday, Wednesday, and Friday) of IHHE (Intermittent Hypoxia-Hyperoxia Exposure) session using the MITOVIT® Hypoxic Training System (COMMIT GmbH, Salzgitter, Germany). They will breathe air with an oxygen concentration (FiO2) ranging from 10-14% for 5 minutes, followed by 3 minutes of rest in hyperoxia (FiO2 30-40%), for a total of 6 cycles. During the hypoxic phase, oxygen saturation will be maintained between 85-92%, while during the hyperoxic phase, it will be kept above 95%. This process is regulated by the device's AI. Participants will be asked to sit and breath normally in each exposure. An attendance checklist will be used to monitor compliance with the intervention
  Interventions: Device: Device: Hypoxic Gas Mixture
- Control group (Sham Comparator): The Sham Group (SG) will follow a 6-week sham intervention protocol with three weekly sessions (Monday, Wednesday, and Friday) of 5 cycles of 6 minutes per session with an FiO2 of 21% using the MITOVIT® Hypoxic Training System (COMMIT GmbH, Salzgitter, Germany). Participants will be asked to sit and breath normally in each exposure. An attendance checklist will be used to monitor compliance with the placebo intervention.
  Interventions: Other: Sham Hypoxic-Hyperoxic exposure

INTERVENTIONS:
Device: Device: Hypoxic Gas Mixture — The EG (Experimental Group) will undergo a 6-week intervention protocol of IHHE (Intermittent Hypoxia-Hyperoxia Exposure) using the MITOVIT® Hypoxic Training System (COMMIT GmbH, Salzgitter, Germany). They will breathe air with an oxygen concentration (FiO2) ranging from 10-14% for 5 minutes, followed by 3 minutes of rest in hyperoxia (FiO2 30-40%), for a total of 6 cycles. During the hypoxic phase, oxygen saturation will be maintained between 85-92%, while during the hyperoxic phase, it will be kept above 95%. This process is regulated by the device's AI. Participants will be asked to sit and breath normally in each exposure. An attendance checklist will be used to monitor compliance with the intervention
  Arms: Intervention group
Other: Sham Hypoxic-Hyperoxic exposure — The Sham Group (SG) will follow a single session protocol of 5 cycles of 6 minutes per session with an FiO2 of 21% using the MITOVIT® Hypoxic Training System (COMMIT GmbH, Salzgitter, Germany). Participants will be asked to sit and breath normally in each exposure. An attendance checklist will be used to monitor compliance with the placebo intervention.
  Arms: Control group

SUMMARY:
The supply of oxygen is essential for energy production, recovery from efforts, and human life. Intermittent Hypoxia-Hyperoxia Exposure (IHHE) is a novel technique in which the subject is exposed to a respiratory environment with reduced oxygen fraction, controlled through a specific software, using a facial mask and a hypoxic generation device. The objective of this study is to determine if there is a relationship between intermittent hypoxia-hyperoxia exposure and cardiorespiratory condition, blood pressure, and arterial oxygen saturation.

According to our hypothesis, acute IHHE in elderly adults may influence cardiorespiratory condition, inflammatory biomarkers, blood pressure, and arterial oxygen saturation.

The study will be conducted as a randomized clinical trial. The subjects will be divided into two groups: the experimental group will undergo an IHHE session, breathing air with an oxygen concentration (FiO2) ranging from 10-14% for 1-5 minutes, with 1-3 minutes of rest in hyperoxia (FiO2 30-40%) for a total of 4-8 cycles, based on their acute response to hypoxia. The sham group will undergo a 5-cycle protocol with an FiO2 of 21%.

Both groups will follow a 6-week protocol with three weekly sessions (Monday, Wednesday, and Friday).

ELIGIBILITY:
Inclusion Criteria:

* Being over 65 years old.
* Having no previous experience in hypoxic training.
* Engaging in less than 150 minutes of physical activity per week.

Exclusion Criteria:

* Having any pathology that prevents the subject from being independent in terms of walking and functionality.
* Subjects with impaired cognitive abilities.
* Subjects with pulmonary hypertension, decompensated heart or respiratory disease.
* To have or have had cancer

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-01-28 (Estimated); Study Completion 2025-02-05 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | 24 hours before intervention and 24 hours after 6 week intervention
  The analysis of Heart Rate Variability will be conducted using a heart rate monitor. Cardiac electrical signals will be monitored with a band placed on the chest for 5 minutes with the subject in supine position on a stretcher, in a quiet environment, soft light, and a comfortable temperature. Subjects are instructed not to speak or make voluntary movements during this analysis.

SECONDARY OUTCOMES:
Blood pressure | 24 hours before intervention and 24 hours after 6 week intervention
  Both systolic and diastolic blood pressure will be assesed using a standard digital sphygmomanometer (Omron HEM-705CP, Omron Healthcare, Inc, Lake Forest, IL)
Arterial oxygen saturation | 24 hours before intervention and 24 hours after 6 week intervention
  Arterial oxygen saturation will be assessed using a device Nonin® 3230 (Nonin Medical, Inc. Plymouth, MN, EEUU)
Respiratory muscle strength | 24 hours before intervention and 24 hours after 6 week intervention
  It will be assessed using a MicroRPM® (MicroMedical, UK).The MicroRPM® is likely a respiratory pressure meter or manometer designed for measuring respiratory muscle strength. It typically includes a mouthpiece connected to a pressure sensor, and the device measures the force or pressure generated during respiratory maneuvers. The person will be instructed to take a maximal deep breath in, and then exhale to residual volume. After that, they will be asked to inhale forcefully against the resistance provided by the MicroRPM®. This measures the strength of the inspiratory muscles. The measures will be expressed in cmH2O.
Pulmonary function | 24 hours before intervention and 24 hours after 6 week intervention
  Pulmonary function tests will be conducted using the Air Smart Spirometer (Pond Healthcare Innovation, Sweden) following the criteria set by the American Thoracic Society (ATS) and the European Respiratory Society (ERS). Measurements included Forced Vital Capacity (FVC) and forced expiratory volume in one second (FEV1), expressed in milliliters, as well as the FEV1/FVC ratio
Inflammatory biomarkers | 24 hours before intervention and 24 hours after 6 week intervention
  C-reactive protein concentration measurements will be taken. A nurse will collect venous blood samples from the antecubital vein after a minimum of 10 hours of overnight fasting. The samples will be centrifuged at 1,800 rpm to extract the serum, which will be stored at -80°C. For analysis, an ELISA microplate reader (SpectraMax PLUS 384, Molecular Devices, San Jose, CA, USA) will be used, following the manufacturer's instructions.

IPD SHARING:
Plan to Share IPD: Yes